CLINICAL TRIAL: NCT04465786
Title: A Closed-loop Brain-computer Interface for Paretic Hand Stimulation After Stroke
Brief Title: A Closed-loop Brain-computer Interface for Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-08-017B
Record Dates: First submitted 2020-04-20; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Stroke; Sensorimotor rhyme; Brain-computer interface
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It may be hard to acquire stable sensorimotor rhythm from the affected motor cortex for patient without a response of paretic hand. A few studies suggest two ways to approaching closed-loop therapy: peripherally extracting the residual signals, for example electromyogram (EMG) at proximal muscles (deltoids) and centrally extracting the activity patterns from unaffected hemisphere during attempting to move paretic hand. Therefore, understanding neural signatures of residual upper extremity movement among stroke patients might help in discovering potential therapeutic target and developing tailored brain-computer interface (BCI) therapy. Additionally, 59.4% of stroke patients in acute stage impair at least one somatosensory modality. It remains unclear whether the patient with somatosensory impairment hinder BCI effect.

DETAILED DESCRIPTION:
Investigators will consecutively enroll subacute (1-4 weeks after stroke onset) patients with first-time, unilateral, subcortical stroke and age-matched healthy controls. All participants will carry on 2 sequential experiments. In the first experiment, participants will perform 2 motor tasks using either paretic/nondominant upper extremity or non-paretic/dominant upper extremity, called motor attempt (M) condition or calibration condition. The second experiment contains 3 conditions: cyclic functional electrical stimulation (cFES), cFES during motor attempt (M-cFES), and functional electrical stimulation during brain-computer interface (BCI-FES) in random order. The sensorimotor oscillations from the electroencephalography (EEG), upper extremity sensorimotor function score (Fugl-Meyer test, Action Research Arm test, and Revised Nottingham Sensation Assessment), corticospinal excitability from the transcranial magnetic stimulation (TMS), and resting-state functional and structural neuroimage from magnetic resonance imaging (MRI) will be assessed before and after the final experiment, as well as 3 months after stroke.

ELIGIBILITY:
Inclusion Criteria:

* first-ever, unilateral infarction or hemorrhage at middle cerebral artery or posterior cerebral artery territory
* early subacute phase of stroke (between 1 and 4 weeks after stroke onset)

Exclusion Criteria:

* electroencephagraphy feature is not usable
* Fugl-Meyer Assessment of Upper Extremity score is over 50
* ataxia
* global aphasia
* concomitant neurological diseases
* psychiatric diseases
* participating in other interventional research during this period
* other conditions might interfere with experiment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized participants and healthy controls will be recruited from the Taipei Veterans General Hospital.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-07-13 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensorimotor rhythms | Baseline, during experimental procedures
  electroencephalography

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | At baseline (1-4 week of stroke) and at 3 months after stroke
  Fugl-Meyer Assessment (FMA) measures both upper-limb and lower-limb motor function. The total score of FMA ranges from 0 to 100, which higher score indicates better motor recovery.
Action Research Arm test | At baseline (1-4 week of stroke) and at 3 months after stroke
  Action Research Arm test (ARAT) measures specific upper-limb and hand function. The total score of ARAT ranges from 0 to 57, which higher score indicates better motor function.
Revised Nottingham Sensation Assessment | At baseline (1-4 week of stroke) and at 3 months after stroke
  Revised Nottingham Sensation Assessment (rNSA) measures various upper-limb sensory function. The total score of rNSA ranges from 0 to 151, which higher score indicates better somatosensory function.
Motor Activity Log | At baseline (1-4 week of stroke) and at 3 months after stroke
  Motor Activity Log (MAL) measures real-use of upper-limb. The averaged index of MAL ranges from 0 to 5, which higher index indicates more frequently use of paretic upper limb.
Resting motor threshold | At baseline (1-4 week of stroke) and at 3 months after stroke
  Transcranial magnetic stimulation test
Motor evoked potential | At baseline (1-4 week of stroke) and at 3 months after stroke
  Transcranial magnetic stimulation test
Resting-state brain connectivity | At baseline (1-4 week of stroke) and at 3 months after stroke
  Magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No